CLINICAL TRIAL: NCT01535508
Title: Open Label Clinical Trial of Vitamin D Dosage Tolerability, and Effect on Behavioral Measures in Children With Autism
Brief Title: Open Label Clinical Trial of Vitamin D in Children With Autism
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VitD11-06899
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Autism; Vitamin D Deficiency
MeSH Terms: conditions — Autistic Disorder; Vitamin D Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liquid Vitamin D (Experimental)
  Interventions: Drug: Liquid Vitamin D

INTERVENTIONS:
Drug: Liquid Vitamin D — 300 IU/Kg/day not to exceed 10,000 IU/day.
  Other Names: Ddrops

SUMMARY:
Primary: to investigate tolerability of interventional high dose Vitamin D3 supplementation, titrated to reach serum levels near the high end of the reference range (30-100 ng/ml), in vitamin D deficient pediatric Autism Spectrum Disorder (ASD) patients.

The study will determine if initial safety and effect estimates predict that a double blind randomized control trial (RCT) with a larger set of patients will be worthwhile in the localization of this treatment aimed at improving the symptoms of ASDs.

Exploratory: to determine efficacy of high dose D3 replacement for improvement in the core symptoms of autism, including sociability, eye contact, anger outbursts, stimming behavior, and sleep, as determined by parental and clinical evaluation scales.

DETAILED DESCRIPTION:
data is still being collected

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism from DSM-IV TR and ADOS
* Moderate but less than severe on CGI-Severity scale
* IQ > 40
* ZRT 25(OH)D blood spot test < 30 ng/ml
* Age 3-8 years old

Exclusion Criteria:

* Developmental delays prior to 12 months of age
* history of head trauma
* seizure in the past year
* bleeding disorder
* history of kidney or liver disease
* clinically significant low white blood cell count
* PDD-NOS, Rett's syndrome, Childhood Disintegrative Disorder or Fragile X syndrome
* current supplementation with Vitamin D, Vitamin A or cod-liver oil

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2012-02; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression Scale - Improvement (CGI-I) | Baseline and 12 weeks from Baseline
  Assessment of global changes in severity of autistic symptoms. CGI-I scores formulated by the clinician based on parent interview of changes in the child's behavior and from direct clinical observation, where scores of 0 = no improvement,1 = minimally improved, 2 = much improved, and 3 = very much improved.

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Hendren, DO, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States